CLINICAL TRIAL: NCT02112721
Title: Can Vitamin D Supplementation Prevent Type 2 Diabetes by Improving Insulin Sensitivity and Secretion in Overweight Humans?
Brief Title: Can Vitamin D Supplementation Prevent Type 2 Diabetes?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: University of Victoria (Other); University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Barbora de Courten, Associate Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1047897
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Group (Experimental): Each participant will be given an initial stat dose of 2500 μg (100,000 IU) of Ostelin (Reckitt Benckiser). Thereafter, participants will take 100 μg/day (4,000 IU, 4 tablets) Ostelin daily for a period of 16 weeks.
  Interventions: Dietary Supplement: Vitamin D
- Placebo group (Placebo Comparator): Each participant will be given an equivalent number of placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Other Names: Ostellin
  Arms: Vitamin D Group
Dietary Supplement: Placebo
  Arms: Placebo group

SUMMARY:
The aim of this study is to determine whether vitamin D supplementation in overweight/obese individuals with vitamin D deficiency can improve insulin secretion and/or insulin resistance by decreasing subclinical inflammation.

Results of the present study may help to identify new strategies to prevent type 2 diabetes in high-risk groups (i.e. overweight and obese individuals, and individuals with a strong family history of diabetes).

Hypothesis: That increasing plasma 25(OH)D concentrations in healthy individuals at risk for type 2 diabetes with low vitamin D levels through vitamin D supplementation, will improve insulin sensitivity and also insulin secretion by reducing the underlying sub-clinical chronic inflammation.

Aims: To establish whether 16-week vitamin D supplementation given to healthy individuals with low vitamin D levels will:

1. improve insulin sensitivity (in vivo and tissue) and/or insulin secretory function
2. determine whether this relationship is mediated by a reduced chronic inflammation

DETAILED DESCRIPTION:
Numerous studies documented that low vitamin D levels are a serious health risk. Despite the sunny climate in Australia, low vitamin D status is becoming increasingly prevalent and people with vitamin deficiency represent more than 30% of the healthy Australian population. Although sun exposure can maintain good vitamin D levels, often sun exposure is limited as people work long hours indoors, and use sunscreen or protective clothing to reduce skin cancer risk when outdoors. Moreover, it is difficult to obtain sufficient vitamin D from food alone; few foods are naturally rich in vitamin D and in Australia, few foods are fortified.

While the importance of vitamin D for bone mineralization is well known, it is less clear how vitamin D protects against type 2 diabetes and cardiovascular disease. Every day in Australia around 275 adults develop diabetes and its prevalence continues to rise.

We are therefore arguing for a well-designed intervention trial to define the preventive potential and physiological mechanisms of the effects of vitamin D supplementation. In addition, we plan to explore the mechanisms underlying the relationship between vitamin D deficiency and the risk for type 2 diabetes, via its influence on chronic inflammation. Our clinical trial will focus on healthy adults with low vitamin D status and will examine the effects on insulin sensitivity and secretion measured by 'gold standard' methodology when vitamin D is restored to optimum levels. It is in particularly important to determine whether vitamin D affects both or only one of these defects because there is evidence from observational studies that there is a relationship between vitamin D levels and both insulin sensitivity and secretion.

The proposed intervention study will potentially supply important evidence on how restoring vitamin D levels may protect against type 2 diabetes. Such findings could have direct relevance for novel approaches to diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 or <60 years,
* 25(OH)D < 50 nmol/L
* Weight change < 5 kg in last 12 months
* BMI >25kg/m2 but weight <159kg due to DEXA scan restrictions
* Non-diabetic, no allergy, non-smoker, no high alcohol use
* No current intake of medications including vitamin supplements
* No kidney, cardiovascular, haematological, respiratory, gastrointestinal, endocrine or central nervous system disease, as well as no psychiatric disorders, no active cancer within the last five years; no presence of acute inflammation (by history, physical or laboratory examination)
* Not menopausal, pregnanct or lactating

Exclusion Criteria:

* Age <18 or > 60 years
* 25(OH)D > 50 nmol/L
* Weight change > 5 kg in last 12 months
* Diabetes (diagnosed or oral glucose tolerance test (OGTT), hypercalcaemia, allergy
* Current smoking habit, high alcohol use
* Current intake of medications including vitamin supplements
* Kidney, cardiovascular, haematological, respiratory, gastrointestinal, endocrine or central nervous system disease, as well as psychiatric disorder, active cancer within the last five years; presence of acute inflammation (by history, physical or laboratory examination)
* Menopause, pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Initial Insulin Sensitivity Measure using Euglycaemic glucose clamp | Week 1
  The clamp will be used to measure insulin sensitivity. The clamp is initiated by an intravenous bolus injection of insulin (9milliUnit/kg). Insulin is then constantly infused at a rate of 40 milliUnit.m-2.min-1 for 120 min into an arm vein, whilst glucose is variably infused to maintain euglycaemia. Plasma glucose values will be monitored every 5 minutes during the clamp and the variable infusion rate of glucose is adjusted to maintain blood glucose at a constant value of 5mmol/L.
Follow up Insulin Sensitivity Measure using Euglycaemic glucose clamp | Week 17
  The clamp will be used to measure insulin sensitivity. The clamp is initiated by an intravenous bolus injection of insulin (9milliUnit/kg). Insulin is then constantly infused at a rate of 40 milliUnit.m-2.min-1 for 120 min into an arm vein, whilst glucose is variably infused to maintain euglycaemia. Plasma glucose values will be monitored every 5 minutes during the clamp and the variable infusion rate of glucose is adjusted to maintain blood glucose at a constant value of 5mmol/L.

SECONDARY OUTCOMES:
Initial measurement of inflammatory markers | Week 1
  Plasma inflammatory markers (interleukin 1β, 6, 8 and 10, TNFα, macrophage migration inhibitory factor, monocyte chemotactic protein-1) will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA) (interassay Coefficients of Variation: 7.2%, 10.2%, 5.8%, respectively). Plasma C- reactive protein (hsCRP) via a high sensitivity assay (BN-II nephelometer; Dade Behring Diagnostics, NSW).
Follow Up Measurement of inflammatory markers | Week 17
  Plasma inflammatory markers (interleukin 1β, 6, 8 and 10, TNFα, macrophage migration inhibitory factor, monocyte chemotactic protein-1) will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA) (interassay Coefficients of Variation: 7.2%, 10.2%, 5.8%, respectively). Plasma C- reactive protein (hsCRP) via a high sensitivity assay (BN-II nephelometer; Dade Behring Diagnostics, NSW).
Initial Measure of Adiposity (DEXA) | Week 1
  body composition by dual energy x-ray absorptiometry (DEXA), which is a non-invasive assessment of soft tissue composition by region with a precision of 4-5%; central adiposity assessed in duplicate using a constant-tension tape for taking waist, and hip circumference. Bioimpedance measurement will be also collected for validation purposes.
Follow Up Measure of Adiposity (DEXA) | Week 17
  body composition by dual energy x-ray absorptiometry (DEXA), which is a non-invasive assessment of soft tissue composition by region with a precision of 4-5%; central adiposity assessed in duplicate using a constant-tension tape for taking waist, and hip circumference. Bioimpedance measurement will be also collected for validation purposes.
Initial Oral Glucose Tolerance Test - OGTT | Week 1
  After a 10-12 h overnight fast, participants will ingest 75g of glucose over 2 mins. Blood samples will be drawn at 0, 30, 60, 90 and 120 min for plasma glucose and insulin concentrations. We will evaluate the area under the curve.
Follow Up Oral Glucose Tolerance Test -OGTT | Week 17
  After a 10-12 h overnight fast, participants will ingest 75g of glucose over 2 mins. Blood samples will be drawn at 0, 30, 60, 90 and 120 min for plasma glucose and insulin concentrations. We will evaluate the area under the curve.
Initial Acute Insulin Secretory Response - Intravenous Glucose Tolerance Test | Week 1
  This will be measured in response to 25g intravenous glucose and calculated as the average incremental plasma insulin level from the third to the fifth minute after the glucose bolus.
Follow up Acute Insulin Secretory Response- Intravenous Glucose Tolerance Test | Week 17
  This will be measured in response to 25g intravenous glucose and calculated as the average incremental plasma insulin level from the third to the fifth minute after the glucose bolus.

OTHER OUTCOMES:
Initial - Other Tissue Analyses | Week 1
  We will measure changes in the expression and activation of important insulin signalling proteins, including the insulin receptor,and we will measure inflammation markers in skeletal, muscle and adipose tissue.
Follow Up- Other Tissue Analyses | Week 17
  We will measure changes in the expression and activation of important insulin signalling proteins, including the insulin receptor,and we will measure inflammation markers in skeletal, muscle and adipose tissue.
Resting systolic and diastolic blood pressure | Week 1
  Resting systolic and diastolic blood pressure and pulse rate will be measured using an automated oscillometric measurement system (Dinamap, USA) after a 30 minute rest.
Follow up Resting systolic and diastolic blood pressure | Week 17
  Resting systolic and diastolic blood pressure and pulse rate will be measured using an automated oscillometric measurement system (Dinamap, USA) after a 30 minute rest.
Initial Arterial waveform measurement | Week 1
  This is done with the BP+ device (Uscom, Australia). This is a device for non-invasive measurement of central blood pressure and augmentation index using an oscillometric method.
Follow up Arterial waveform measurement | Week 17
  This is done with the BP+ device (Uscom, Australia). This is a device for non-invasive measurement of central blood pressure and augmentation index using an oscillometric method.
Initial Beck Depression Inventory | Week 1
  The Beck Depression Inventory (BDI), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. It is designed for individuals aged 13 and over, and is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex.
Follow Up Beck Depression Inventory | Week 17
  The Beck Depression Inventory (BDI), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. It is designed for individuals aged 13 and over, and is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex.
Initial Pain Impact Questionnaire (PIQ-6 questionnaire) | Week 1
  PIQ-6 measures the severity of pain and its impact on work and leisure activities, as well as on emotional well-being within a variety of diseases and general populations. This survey is intended for adults 18 years of age and older.
Follow Up Pain Impact Questionnaire (PIQ-6 questionnaire) | Week 17
  PIQ-6 measures the severity of pain and its impact on work and leisure activities, as well as on emotional well-being within a variety of diseases and general populations. This survey is intended for adults 18 years of age and older.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora de Courten, PhD, MD, Principal Investigator — Monash University
Locations (1):
- Monash Centre for Health Research and Implementation, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Stark R, Feehan J, Mousa A, Andrews ZB, de Courten B. Liver-expressed antimicrobial peptide 2 is associated with improved pancreatic insulin secretion in adults with overweight and obesity. Diabetes Obes Metab. 2023 May;25(5):1213-1220. doi: 10.1111/dom.14968. Epub 2023 Jan 19. PMID 36597795
- [Derived] Mousa A, Naderpoor N, Wilson K, Plebanski M, de Courten MPJ, Scragg R, de Courten B. Vitamin D supplementation increases adipokine concentrations in overweight or obese adults. Eur J Nutr. 2020 Feb;59(1):195-204. doi: 10.1007/s00394-019-01899-5. Epub 2019 Jan 16. PMID 30649593
- [Derived] Scott D, Mousa A, Naderpoor N, de Courten MPJ, Scragg R, de Courten B. Vitamin D supplementation improves waist-to-hip ratio and fasting blood glucose in vitamin D deficient, overweight or obese Asians: A pilot secondary analysis of a randomised controlled trial. J Steroid Biochem Mol Biol. 2019 Feb;186:136-141. doi: 10.1016/j.jsbmb.2018.10.006. Epub 2018 Oct 12. PMID 30321667
- [Derived] Mousa A, Naderpoor N, de Courten MP, Teede H, Kellow N, Walker K, Scragg R, de Courten B. Vitamin D supplementation has no effect on insulin sensitivity or secretion in vitamin D-deficient, overweight or obese adults: a randomized placebo-controlled trial. Am J Clin Nutr. 2017 Jun;105(6):1372-1381. doi: 10.3945/ajcn.117.152736. Epub 2017 May 10. PMID 28490514
- [Derived] de Courten B, Mousa A, Naderpoor N, Teede H, de Courten MP, Scragg R. Vitamin D supplementation for the prevention of type 2 diabetes in overweight adults: study protocol for a randomized controlled trial. Trials. 2015 Aug 7;16:335. doi: 10.1186/s13063-015-0851-6. PMID 26246241